**Project Title:** Public Support for Prison Nutrition Standards

ClinicalTrials.gov ID: NCT06840600

**Date:** 3/26/25

# CTGov Analytic plan

**Title:** Public Support for Prison Nutrition Standards

**NCT #:** NCT06840600

### <u>Introduction</u>

This study focuses on public support for prison nutrition standards—a policy that would require U.S. prisons to serve meals that abide by the USDA Dietary Guidelines for Americans. Specifically, we aim to examine whether different framings explaining the rationale for the policy change public support for prison nutrition standards. The study will also explore whether demographic characteristics, such as political affiliation or previous interaction with the criminal legal system moderate the effect of policy rationale on public support. This document pre-specifies our planned analytic approach prior to data collection.

### Study protocol

In an online survey, participants will be asked to imagine a new U.S. policy which would require prisons to serve meals that meet the government definition of healthy. In a between-subjects experiment, participants will be randomly assigned to view 1 of 3 different rationales for the new policy—public safety, right-to-health, or cost-saving—or be assigned to a control arm where no rationale is given. After viewing the rationale, participants will be asked whether they would strongly support, somewhat support, neither support or oppose, somewhat oppose, or strongly oppose the policy. Participants will also answer demographic questions.

### Statistical analysis plan

#### **Predictions**

We predict that public support will be higher among participants who are assigned any of the 3 policy rationales vs. no rationale (control). We do not have predictions as to which rationale will elicit the highest public support.

#### Statistical methods

Using linear regression, we will regress policy support on indicator variables for the experimental arm, excluding the control arm as referent. In this model, policy support will be treated as a continuous variable with responses ranging from 1 (representing strongly oppose) to 5 (strongly support). Analyses will estimate average differential effects (ADE, differences in predicted means) for each rationale compared to the control. We will use a two-sided critical alpha of 0.05 to conduct all statistical tests. All confidence intervals presented will use a 95% confidence level. We will then use pairwise comparisons to compare the predicted outcomes for each rationale to one another, using Bonferroni-Holm corrected p-values, to adjust for these 3 additional post-hoc tests.

We will use linear regression to examine correlates of policy support. We will regress policy support on the following demographic characteristics in a multivariable model:

- Reason for policy (experimental arm, with control arm as referent)
- Age
- Gender
- Race/ ethnicity
- Income
- Education
- Political party affiliation
- Having prior interactions with the criminal legal system
- Holding biases toward people who are incarcerated

For all analyses, we will exclude participants who complete <90% of the survey or who complete the survey implausibly quickly (defined as <1/3 of the median completion time).

## Sample size needs

This study will occur as an auxiliary study to an experiment examining the impact of nudges on improving the healthfulness and environmental sustainability of grocery purchases (i.e., the parent study). The total sample size (~1,200 participants) was calculated based on the anticipated effect sizes in the parent study.